CLINICAL TRIAL: NCT05048290
Title: Building a Diverse Biomedical Workforce Through Communication Across Difference
Brief Title: Communication Skills to Build a Diverse Biomedical Workforce
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: PI Request
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 2019-1010; NCI-2020-04436 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2019-1010 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2021-09-08; First posted 2021-09-17 (Actual); Last update posted 2025-06-11 (Actual); Status verified 2025-06

CONDITIONS: Behavioral Disorder
MeSH Terms: conditions — Mental Disorders | interventions — Early Intervention, Educational; Educational Status; Methods

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group I (communication workshops, video, surveys) (Experimental): Participants complete 2 communication workshops about conversational skills and development of a video about the summer student's research experience over 3 hours each during the second week of the summer research experience and 2-3 weeks before the conclusion of summer experience. Participants also complete surveys over 15 minutes each about their communication, their engagement with research, mentoring experience, and current career intentions, before participating in the workshop, after the second workshop and at 6 months after the conclusion of the summer experience.
  Interventions: Other: Communication Skills Training; Other: Educational Intervention; Other: Survey Administration
- Group II (generic communication workshops, surveys) (Active Comparator): Participants complete 2 generic communication workshops about networking and presentation skills over 3 hours each during the second week of the summer experience and 2-3 weeks before the conclusion of summer experience. Participants also complete surveys over 15 minutes each about their communication, their engagement with research, mentoring experience, and current career intentions, before participating in the workshop, after the second workshop and at 6 months after the conclusion of the summer experience.
  Interventions: Other: Communication Skills Training; Other: Survey Administration

INTERVENTIONS:
Other: Communication Skills Training — Participate in communication workshops
  Arms: Group I (communication workshops, video, surveys)
Other: Communication Skills Training — Participate in generic communication skills workshops
  Arms: Group II (generic communication workshops, surveys)
Other: Educational Intervention — Develop a video
  Other Names: Education for Intervention; Intervention by Education; Intervention through Education; Intervention, Educational
  Arms: Group I (communication workshops, video, surveys)
Other: Survey Administration — Complete surveys

SUMMARY:
This trial investigates how receiving instruction in communication skills affects short and long-term career outcomes for students, postdoctoral fellows, and future faculty. This may help researchers learn more about the factors that may help or block career goals and career persistence of trainees.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Determine communication across difference (CAD) workshop effects over time using experimental and control dyads of summer students and their matched junior mentors.

Ia. Develop and deliver CAD skills workshops to dyads of students and junior mentors.

Ib. Test CAD workshop effects for individual participants with pre-, post-, and follow-up surveys of model variables over the course of the intervention.

II. Identify causal relationships of the social-influence variables with experimental and control groups of dyads over the 9-month course of the intervention.

IIa. Assess the psychological processes and causal relationships for students linking CAD to career intentions.

IIb. Assess the psychological processes and causal relationships for junior mentors linking CAD to career intentions and intentions to mentor diverse students in the future.

IIc. Assess the paired interaction effects between dyad members using pre-, post-, and follow-up model variables over the course of the intervention.

III. Assess long-term outcomes of the intervention and predictive utility of the student and mentor models by measuring changes in Hallmarks of Success: distal career persistence and network growth for students and junior mentors, as well as junior mentors' engagement in mentoring of diverse students.

OUTLINE: Dyads of summer students and their matched junior mentors are assigned to 1 of 2 groups.

GROUP I (EXPERIMENTAL): Participants complete 2 communication workshops about conversational skills and development of a video about the summer student's research experience over 3 hours each during the second week of the summer research experience and 2-3 weeks before the conclusion of summer experience. Participants also complete surveys over 15 minutes each about their communication, their engagement with research, mentoring experience, and current career intentions, before participating in the workshop, after the second workshop and at 6 months after the conclusion of the summer experience.

GROUP II (CONTROL): Participants complete 2 generic communication workshops about networking and presentation skills over 3 hours each during the second week of the summer experience and 2-3 weeks before the conclusion of summer experience. Participants also complete surveys over 15 minutes each about their communication, their engagement with research, mentoring experience, and current career intentions, before participating in the workshop, after the second workshop and at 6 months after the conclusion of the summer experience.

ELIGIBILITY:
Inclusion Criteria:

* FOR SUMMER STUDENTS: Currently an undergraduate, medical student, or early Master's or Doctor of Philosophy (PhD) level student who is participating in a structured summer research program and receiving daily research supervision from a junior mentor (defined as a Master's or PhD level graduate student, a postdoctoral fellow, or an instructor) within a faculty member's research team
* FOR JUNIOR MENTORS: Currently a Master's or PhD student; postdoctoral trainee; or instructor working within a faculty member's research team and supervising a summer research student

Exclusion Criteria:

* FOR SUMMER STUDENTS: High school students

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-05-19 (Actual); Primary Completion 2024-12-30 (Actual); Study Completion 2024-12-30 (Actual)

PRIMARY OUTCOMES:
Degree completion rates | Through study completion, an average of 1 year
  Will be assessed in both summer students and junior mentors.

CONTACTS AND LOCATIONS:
Overall Officials: Carrie Cameron, Principal Investigator — M.D. Anderson Cancer Center

REFERENCES:
- See also: M.D. Anderson Cancer Center — http://www.mdanderson.org

DOCUMENTS (1):
  • Informed Consent Form (2023-01-06): https://cdn.clinicaltrials.gov/large-docs/90/NCT05048290/ICF_000.pdf